CLINICAL TRIAL: NCT04252508
Title: Impact of a Double-reading Animated Film (Child, Parents) in Preoperative on the Anxiety of Children Upon Arrival at the Operating Room
Acronym: VERAPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2018/57
Record Dates: First submitted 2019-10-15; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-10

CONDITIONS: Anxiety; Surgery; Pediatric ALL
Keywords: Preoperative- Child; Double-reading movie
MeSH Terms: conditions — Anxiety Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With animated film (Experimental): An animated film depicts the child and the caregivers in the form of avatars and retraces his journey from his room to the transfer area, then to the the operating room and finally to the post-intervention ward.
  Interventions: Other: Animated film
- Standard route (No Intervention): The information about the surgery will be given by the surgeon during the consultation.
  Those about anaesthesia will be delivered by anaesthesiologist during the anaesthetic consultation.

INTERVENTIONS:
Other: Animated film — An animated film depicts the child and the caregivers in the form of avatars and retraces his journey from his room to the transfer area, then to the the operating room and finally to the post-intervention ward.
  Arms: With animated film

SUMMARY:
Preoperative anxiety affects 40 to 60% of children. A literature review concluded that effective preparation strategies must involve parents, must be appropriate to their age and proposed upstream of the intervention.

A double-readinganimated film aimed at informative was created for the children and their parents/legal guardians in order to solve the problem of anxiety found at the arrival of children in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Child boy or girl.
* 3 to 7 years old.
* programmed for: removal of tonsils, vegetations, paracentesis or installation of trans-tympanic aerators, pre-heliceal fistula, otoplasty, myringoplasty
* Scheduled intervention in the outpatient department of specialized surgeries or hospitalization of a postoperative night.
* Accompanied by an adult, French-speaking, whose child lives at home.
* Of which the holders of the parental authority formulated their non-opposition to the participation of their child and gave their signed agreement for the realization of videos of their child.
* Assent of the child for children aged 6 to 7
* Parents affiliated to social security

For the group under study only:

- Support available at home that can watch the movie on the internet

Exclusion Criteria:

* Child having already had surgery.
* Presence of associated disability (blindness, profound deafness, autistic disorders).
* Child having anxiolytic treatment.
* Child to be operated within less than 2 days

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-04-09 (Estimated); Study Completion 2021-04-09 (Estimated)

PRIMARY OUTCOMES:
the child's anxiety score obtained from the M-Ypass scale at the time of induction in the operating room. | The duration of this visit will be about 3 hours, between the reception at the outpatient and the time of induction in intervention room, end of the study
  Evaluation of this outcome measure will be made between 0 and 6 months after the inclusion. m-Ypass scale (Modified Yale Preoperative Anxiety Scale), a hetero-evaluation scale, is designed to assess preoperative anxiety in children aged 3 to 7 years.
  It has 18 items divided into 4 groups (activity, vocalizations, emotional expression, apparent state of awakening). Each group having a different number of items (4 or 6), quotients are calculated and then added together to obtain a total score ranging from 0 to 100 (Appendix 2: Anxiety score of Yale Mulhouse and Colmar).
  The children will be filmed at 3 times of their care on the day of the intervention.
  The reading of these videos will be done afterwards by two nurses from the Department of Pain Support Unit (CHU Bordeaux, neuroscience center), independent of the services concerned by the study, trained on a scale by the investigator, in order to establish anxiety scores.

SECONDARY OUTCOMES:
the child's anxiety score obtained from the M-Ypass scale | at their arrival in ambulatory service.
  m-Ypass scale (Modified Yale Preoperative Anxiety Scale), a hetero-evaluation scale, is designed to assess preoperative anxiety in children aged 3 to 7 years.
  It has 18 items divided into 4 groups (activity, vocalizations, emotional expression, apparent state of awakening). Each group having a different number of items (4 or 6), quotients are calculated and then added together to obtain a total score ranging from 0 to 100 (Appendix 2: Anxiety score of Yale Mulhouse and Colmar).
  The children will be filmed at 3 times of their care on the day of the intervention.
  The reading of these videos will be done afterwards by two nurses from the Department of Pain Support Unit (CHU Bordeaux, neuroscience center), independent of the services concerned by the study, trained on a scale by the investigator, in order to establish anxiety scores.
the child's anxiety score obtained from the M-Ypass scale at their arrival in ambulatory service | The duration of this visit will be about 3 hours, between the reception at the outpatient and the time of induction in intervention room, end of the study
  Evaluation of this outcome measure will be made between 0 and 6 months after the inclusion. m-Ypass scale (Modified Yale Preoperative Anxiety Scale), a hetero-evaluation scale, is designed to assess preoperative anxiety in children aged 3 to 7 years.
  It has 18 items divided into 4 groups (activity, vocalizations, emotional expression, apparent state of awakening). Each group having a different number of items (4 or 6), quotients are calculated and then added together to obtain a total score ranging from 0 to 100 (Appendix 2: Anxiety score of Yale Mulhouse and Colmar).
  The children will be filmed at 3 times of their care on the day of the intervention.
  The reading of these videos will be done afterwards by two nurses from the Department of Pain Support Unit (CHU Bordeaux, neuroscience center), independent of the services concerned by the study, trained on a scale by the investigator, in order to establish anxiety scores.
the child's anxiety score obtained from the M-Ypass scale | at their arrival at the transfer area of the operating room
  m-Ypass scale (Modified Yale Preoperative Anxiety Scale), a hetero-evaluation scale, is designed to assess preoperative anxiety in children aged 3 to 7 years.
  It has 18 items divided into 4 groups (activity, vocalizations, emotional expression, apparent state of awakening). Each group having a different number of items (4 or 6), quotients are calculated and then added together to obtain a total score ranging from 0 to 100 (Appendix 2: Anxiety score of Yale Mulhouse and Colmar).
  The children will be filmed at 3 times of their care on the day of the intervention.
  The reading of these videos will be done afterwards by two nurses from the Department of Pain Support Unit (CHU Bordeaux, neuroscience center), independent of the services concerned by the study, trained on a scale by the investigator, in order to establish anxiety scores.
the child's anxiety score obtained from the EVA-A for the parent/legal guardian. | at the time of induction in the operating room
  The EVA-A (Numerical Scale for Anxiety) is a self-assessment scale that assesses situational anxiety.
  The question formulated by the professional who makes the welcome interview to the SAS transfer from the operating room to the accompanying person will be the following:
  "Can you on a scale of 0 to 10, evaluate your apprehension? " This will allow an estimate of anxiety between 0 and 10. 0 = no anxiety, 10 = maximum anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Plateau technique Centre François-Xavier Michelet, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No